CLINICAL TRIAL: NCT05093907
Title: An Open-label, Single Center, Phase I/II Clinical Trial to Assess the Maximum Tolerated Dose, Safety and Efficacy of BEY1107 in Combination with Capecitabine in Patients with Metastatic Colorectal Cancer Refractory or Intolerant to Standard of Care
Brief Title: A Study to Evaluate Safety and Efficacy of BEY1107 in Combination with Capecitabine in Patients with Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeyondBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BEY-2021-01
Record Dates: First submitted 2021-09-16; First posted 2021-10-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BEY1107 + Capecitabine (Experimental): Administer BEY1107 in combination with Capecitabine, 3-weeks as 1 cycle.
  Interventions: Drug: BEY1107; Combination Product: Capecitabine

INTERVENTIONS:
Drug: BEY1107 — Administer once daily, PO, 3-week continuous dose.
Combination Product: Capecitabine — Administer twice daily, PO, 2-week continuous dose, followed by 1-week rest period.

SUMMARY:
This is a Phase 1/2 study to evaluate the maximum tolerated dose, safety and efficacy of BEY1107 in combination with capecitabine in patients with metastatic colorectal cancer refractory or intolerant to standard of care (SoC).

DETAILED DESCRIPTION:
In Phase 1, patients who experienced treatment failure of colorectal cancer with the second-line or beyond standard chemotherapy will be enrolled at each dose level of BEY1107 in combination with Capecitabine. Phase 2 will be conducted after RP2D is determined on the Phase 1 results.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged over 19 years or older at the time of Informed Consent.
2. Histopathologically or cytologically diagnosed with colorectal cancer.
3. Patients with unresectable metastatic lesion(s).
4. Patients who experienced treatment failure of colorectal cancer with the second-line or beyond standard chemotherapy (including fluoropyrimidine, oxaliplatin and irinotecan).
5. Subjects who have at least one measurable or evaluable lesion as per RECIST v1.1.
6. Subjects with ECOG performance status 0 or 1.
7. Women of childbearing potential who are not surgically sterile must consent to practice acceptable contraception until 6 months after the end of IP administration and also have the evidence of not being fertile.
8. Non-vasectomized men who consent to use an acceptable contraception by one-self and the partner until 3 months after the end of IP administration.
9. Patients who are fully informed of this trial, voluntarily decide to participate in the trial and provide written consent to comply with requirements for the trial.

Exclusion Criteria:

1. Patients who received radiation therapy, chemotherapy or biological agent including hormone therapy recently.
2. Subjects who had a surgery with general anesthesia within 4 weeks of screening.
3. Subjects with symptomatic brain metastasis.
4. Subjects with peripheral neuropathy.
5. Subjects who had findings of affecting absorptin of the IP with gastrointestinal surgery or impossible oral drug administration.
6. Subjects with systemic disease not suitable for anticancer agent administration at the discretion of the investigator.
7. Subjects who had a cardiovascular disease as of screening.
8. Subjects with history of malignancy other than basal cell carcinoma of the skin or cervical carcinoma in situ or papillary thyroid cancer appropriately treated within 5 years.
9. Gastrointestinal bleeding or ulcer.
10. Dihydro-Pyridine Dehydrogenase (DPD) deficiency.
11. Galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
12. Hypersensitivity to the ingredient(s) of the investigational product (BEY 1107) or capecitabine, 5-FU (fluorouracil).
13. HIV Positive.
14. Ineligible result of HBV, HCV by the investigator.
15. Acute or severe infection.
16. Subjects who take a Sorivudine or brivudine in combination.
17. Subjects who take a combination of tegafur, gimeracil and oteracil potassium or discontinue within 7 days at the screening.
18. Subjects who take a Rifampin and azole class antifungal drugs in combination.
19. Subjects who has labortory findings of inadequate bone marrow, kidney and liver function.
20. Pregnant women, breastfeeding women, or positive findings on the pregnancy test at screening.
21. Subjects with life expectancy of less than 12 weeks by the investigator.
22. Subjects who had been administered other IP within 4 weeks prior to screening.
23. Subjects determined by the investigator to be ineligible for participation in this trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD) assessed by investigator following administration of BEY1107 in combination with Capecitabine | From baseline up to disease progression, approximately 54 weeks
  MTD will be assessed based on adverse events(including DLT assessment), vital signs, 12-lead ECG, laboratory tests, etc.
Objective Response Rate(ORR)(Phase 2) assessed by investigator following administration of BEY1107 in combination with Capecitabine | From baseline up to disease progression, approximately 54 weeks
  ORR defined as proportion of subjects with a overall response of CR or PR

SECONDARY OUTCOMES:
Pharmacokinetic(PK) of Maximum Serum Concentration (Cmax) of BEY1107 in combination with Capecitabine | From baseline up to 24 hour post-dose
  Plasma concentrations at each time point and PK parameters Cmax of BEY1107 will be assessed in the PK sampling cohort
Pharmacokinetic of Time to Reach Maximum Serum Concentration (Tmax) of BEY1107 in combination with Capecitabine | From baseline up to 24 hour post-dose
  Plasma concentrations at each time point and PK parameters Tmax of BEY1107 will be assessed in the PK sampling cohort
Pharmacokinetic of Area Under the Serum Concentration-Time Curve Up to Last Quantifiable Time (AUClast) of BEY1107 in combination with Capecitabine | From baseline up to 24 hour post-dose
  Plasma concentrations at each time point and PK parameters AUClast of BEY1107 will be assessed in the PK sampling cohort
Progression-free survival(PFS) assessed by investigator following administration of BEY1107 in combination with Capecitabine | From baseline up to disease progression, approximately 24 months
  PFS is defined as the time from the start of study treatment to the date of the first documentation of objective PD or death due to any cause, whichever is earlier
Disease control rate(DCR) assessed by investigator following administration of BEY1107 in combination with Capecitabine | From baseline up to approximately 24 months
  DCR is defined as the proportion of participants who achieved a confirmed best overall response (BOR) of complete response (CR), partial response (PR), or stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospial, Seoul, Jongro-go, South Korea